CLINICAL TRIAL: NCT02324127
Title: Clinical Trial of Quantitative Detection Kit for Hsp90α in Hepatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Protgen Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: hsp90a2011-05
Record Dates: First submitted 2014-12-14; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- liver cancer (Experimental): Detect plasma Hsp90α concentration of liver cancer patients
  Interventions: Device: hsp90

INTERVENTIONS:
Device: hsp90 — Detect plasma Hsp90α concentration of lung cancer patients
  Other Names: biomarker

SUMMARY:
Detect plasma Hsp90α concentration of liver cancer patients, healthy volunteers, benign liver diseases.

DETAILED DESCRIPTION:
Detect plasma Hsp90α concentration of liver cancer patients, healthy volunteers, benign liver diseases, validate accuracy, specificity and sensitivity of Hsp90α kit.

ELIGIBILITY:
Inclusion Criteria:

* Liver cancer patients
* Healthy volunteers,
* Benign liver diseases patients

Exclusion Criteria:

* Patients who Previously accepted radiotherapy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Hsp90α Concentration of plasma | 4 months
  Detect Hsp90α Concentration(ng/ml) of plasma and calculate the accuracy, specificity and sensitivity of Hsp90α kit

CONTACTS AND LOCATIONS:
Overall Officials: Shusen Zhen, MD, Principal Investigator — The first hospital of Zhejiang province
Locations (1):
- Zhejiang Medical University Cancer Institute and Hospital, Hangzhou, Zhejiang, China